CLINICAL TRIAL: NCT06560138
Title: An Open-label, Multi-center Phase I Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of SHR-4602 in Subjects With HER2-expressing or HER2-mutated Locally Advanced or Metastatic Solid Tumors
Brief Title: A Trial of SHR-4602 Infusion in Patients With SHR-4602 in Subjects With HER2-expressing or HER2-mutated Locally Advanced or Metastatic Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: In accordance with the strategic decision of the company's senior management team, no participants have been consented or enrolled.
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4602-102
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-09

CONDITIONS: HER2-expressing or HER2-mutated Locally or Metastatic Solid Tumors

STUDY DESIGN:
Intervention Model Description: SHR-4602 injection only
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-4602 Dose level 1 : 2.0 mg/kg, Dose level 2 : 2.5mg/kg (Experimental)
  Interventions: Drug: SHR-4602

INTERVENTIONS:
Drug: SHR-4602 — SHR-4602 will be administered through IV infusion.

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR-4602 in subjects with HER2-expressing or HER2-mutated locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, voluntarily participate in the trial.
2. ECOG PS score 0 or 1
3. Life expectancy ≥ 12 weeks
4. Adequate bone marrow and other vital organ functions
5. Adequate liver function tests
6. HER 2 exprission advanced solid tumor

Exclusion Criteria:

Inclusion Criteria

1. Ability to understand the trial procedures and possible adverse events, voluntarily participate in the trial.
2. ECOG PS score 0 or 1
3. Life expectancy ≥ 12 weeks
4. Adequate bone marrow and other vital organ functions
5. Adequate liver function tests
6. HER 2 exprission advanced solid tumor

Exclusion Criteria

1. Active brain metastases, carcinomatous meningitis/leptomeningeal metastases.
2. Have received surgery (eg. major surgerical treatment for cancer), chemotherapy, molecular targeted therapy, immunotherapy, cell therapy, or radiotherapy within 4 weeks prior to the first dose of investigational drug (palliative radiotherapy within 2 weeks prior to the first dose).
3. Participated in another clinical study with the last dose of study drug received in less than 4 weeks prior to the first dose.
4. Subjects with toxicities and/or complications from prior treatment not recovered to NCI-CTCAE Grade ≤ 1.
5. History of pleural fluid, ascites, or pericardial effusion requiring intervention within 2 weeks prior to the first dose.
6. History of active autoimmune diseases.
7. History of hereditary or acquired bleeding disorders or thrombotic tendency
8. Active hepatitis B (defined as hepatitis B virus surface antigen [HBsAg] positive and serum HBV-DNA copy ≥ 500 IU/mL), hepatitis C
9. History of severe infection within the past 30 days, including but not limited to bacteremia, severe sepsis, pneumonia requiring hospitalization
10. Other malignancies currently or within the past 5 years, except for cured cervical carcinoma in situ
11. Allergy to any component or excipient of the SHR-4602 product,
12. History of severe medical, psychiatric, or social conditions deemed by the investigator to be likely to interfere with a subject's ability to understand, consent, cooperate and participate in the study.
13. Patients with Grade≥2 peripheral neuropathy, except for those with mild symptoms that do not require treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-14 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
the phase II dose (RP2D) of SHR-4602 | From the time when the subjects sign the informed consent form to 45(±3) days after the last dose of SHR-4602, or the start of new anti-tumor treatment (whichever comes first).assessed for a maximum duration of up to 1 year
  RP2D is defined as the dose of SHR-4602 recommended for efficacy study in Phase II. It will be the dose with promising clinical responses observed in the subjects, well tolerated by subjects without exceeding a pre-set number of adverse events.

SECONDARY OUTCOMES:
Cmax | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  Cmax are the maximum observed plasma concentrations of SHR-4602, total antibodies, and free toxin after the first dose, directly observed from data.
Tmax | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  Tmax is the time point when Cmax is observed.
Css, max, | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  Css, max are steady-state maximum concentrations of SHR-4602, total antibodies, and free toxin during multiple dosing, and are directly observed from data.
Css, min | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  Css, min are the steady-state trough concentrations of SHR-4602, total antibodies, and free toxin during multiple dosing, and are directly observed from data.
AUC0-t | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  AUC0-t are the areas under the drug concentration-time curve of SHR-4602, total antibodies, and free toxin from time 0 to the last measurable concentration time point
AUC0-∞ | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  AUC0-∞ are the areas under the drug concentration-time curve of SHR-4602, total antibodies, and free toxin (ER300) from time 0 to infinity
AUCτ | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  AUCτ are the areas under the drug concentration-time curve of SHR-4602, total antibodies, and free toxin between two doses of SHR-4602 after multiple administrations.
t1/2 | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  t1/2 is he elimination half-life
CL | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  CL is the clearance
Vss | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  Vss is volume of distribution
MRT | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  MRT is the mean residence time, of SHR-4602, total antibodies, or free toxin. Those values are calculated using the non-compartmental model.
Rac | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  Rac is the accumulation ratios of SHR-4602, total antibodies, or free toxin. It will be evaluated based on the ratio of exposure following multiple administrations to the single administration
anti-SHR-4602 antibody (ADA) | Pre-set time points: from C1D1 within 1 hour pre-dose to 30 ± 7 days, after EOT up to 1 year
  Approximately 4 mL of blood samples will be collected at pre-set time points and used for immunogenicity-related studies, which may include designation of in-study cut-points, analysis of anti-drug antibody (ADA) and neutralizing antibody, and target interference studies. All ADA assay results obtained will be listed. Samples positive for ADA will be analyzed for titers. The percentage of ADA positive subjects, time to ADA onset, ADA duration will be summarized by dose group.
Objective Response Rate (ORR) | From the first date with measurable disease meeting the CR or PR criteria, to the date of PD or death from any cause, whichever occurs first. assessed for a maximum duration of up to 3 years
  ORR refers to the proportion of subjects with a best overall response of Complete/Partial Response (CR or PR) in subjects with measurable diseases by tumor imaging per RECIST v1.1. For subjects with CR or PR at the first evaluation, the efficacy should be confirmed 4 weeks later or at the next tumor imaging evaluation.
Duration of Response (DoR) | From the first date with measurable disease meeting the CR or PR criteria, to the date of PD or death from any cause, whichever occurs first. assessed for a maximum duration of up to 3 years
  DOR refers to the time from the first occurrence of CR or PR to Progression of Disease (PD) or death from any cause, whichever occurs first, in subjects with objective response. If the subject does not experience PD or death or is lost to follow-up at the end of study, DOR will be censored at the time of the last tumor evaluation. DOR will be estimated using the method of Kaplan-Meier
Disease Control Rate (DCR) | From the first date with measurable disease meeting the CR, PR or SD criteria, to the date of PD or death from any cause, whichever occurs first. assessed for a maximum duration of up to 3 years.
  DCR refers to the proportion of subjects with a best overall response of CR, PR, or Stable Disease (SD). Subjects evaluated as SD should meet the criteria for SD at least once at a minimum of 6 weeks after enrolment.
Progression Free Survival (PFS) | From the first dose of SHR-4602 to the first PD or death from any cause (whichever occurs first). assessed for a maximum duration of up to 3 years
  PFS refers to the time from the first dose of SHR-4602 to the first PD or death from any cause (whichever occurs first) as assessed by the investigator. If the subject does not experience PD or death or receives other anti-tumor treatments at the end of study, PFS will be censored on the date of the last tumor assessment. PFS will also be estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Scientia Clinical Research Limited, Randwick, New South Wales
  - Macquarie University, Sydney, New South Wales
  - Icon Cancer Centre South Brisbane, Brisbane, Queensland
  - Cancer Research SA, Adelaide, South Australia
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria